CLINICAL TRIAL: NCT00933465
Title: Single Blinded Randomised Cross-over Study of Imodium Tablets Versus Imodium Syrup for the Treatment of Faecal Incontinence
Brief Title: Imodium Syrup Versus Imodium Tablets for Faecal Incontinence
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other)
Responsible Party: Miss Karen Nugent, Southampton University hospital NHS trust
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RHMMED0874; eudraCT number; 2009-013776-49
Record Dates: First submitted 2009-07-03; First posted 2009-07-07 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Fecal Incontinence
Keywords: Fecal incontinence
MeSH Terms: conditions — Fecal Incontinence | interventions — Loperamide; Tablets

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tablets first followed by syrup (Experimental): first 6 weeks of study using tablets, then followed by assessment, and then the next 6 weeks using syrup, followed by assessment
  Interventions: Drug: Imodium (Loperamide Hydrochloride) syrup; Drug: Imodium (Loperamide hydrochloride) tablets
- Syrup first followed by tablets (Experimental): first 6 weeks of study using syrup, then followed by assessment, and then the next 6 weeks using tablets, followed by assessment
  Interventions: Drug: Imodium (Loperamide Hydrochloride) syrup; Drug: Imodium (Loperamide hydrochloride) tablets

INTERVENTIONS:
Drug: Imodium (Loperamide Hydrochloride) syrup — syrup (orally), max dose per day; 16x 5ml spoonfuls (80ml) Titrated from low dose to clinically relevant dose as described by the patient and their symptoms.
  Taken at times suitable for the patient, either at regular intervals as defined by patient needs, or as single dose when needed the most.
Drug: Imodium (Loperamide hydrochloride) tablets — tablets (orally) max dose per day; in chronic diarrhea, 8 capsules (16 mg) titrated from low dose to clinically relevant dose as described by patient and their symptoms.
  Taken at times suitable for the patient, either at regular intervals as defined by patient needs, or as single dose when needed the most

SUMMARY:
Faecal incontinence (FI) is a debilitating and often neglected problem. It can be defined as the loss of voluntary control of liquid or solid stool.It is estimated that 2-3% of western adults suffer from FI with prevalence increasing with age, further to this up to 50% of nursing home residents suffer too with it more common in females. Aetiology is often multi-factoral, where obstetric anal sphincter injury is most common is females and iatrogenic anal sphincter injury is most common in males.

Loperamide (imodium) is a constipating agent used as first choice pharmacological agent due to its high efficacy. Trials have suggested it thickens stool consistency and may raise resting anal sphincter pressure, associated with improved clinical function with a reduction in bowel frequency and urgency, a reduction in incontinence and less need for pads.

Loperamide is well tolerated but has been known to cause side effects of abdominal pain and distension, nausea and vomiting and constipation.

Imodium can be taken in two ways; as syrup (1mg/5mls) or tablets (2mg). There have been no comparative studies. Side effects are mainly seen with the tablet form and so it is hypothesized that the syrup form is better tolerated because it is more accurately titrated to effect.

This is a NHS funded single blinded, randomised, cross-over study to assess the clinical effects of Imodium, in tablet and syrup form, on patients presenting with faecal incontinence. Each subject will act as their own control. Patients will be recruited through out-patient visits for their FI, where they will be made aware of the trial. During the trial they will be asked to fill out FI scoring questionnaires and quality of life scores. Also they will undertake two assessments of anal physiology testing squeeze pressures, sensation and compliance at baseline and at the end after three months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 75
* Severe faecal incontinence defined as greater than one episode per week of involuntary loss of either solid or liquid stool as demonstrated by means of a baseline bowel habit and a Vaizey score of greater than 4.
* Competent and willing to fill in questionnaires and attend follow up clinics through out the study period.

Exclusion Criteria:

* Alternating bowel habit, associated with symptoms of constipation. Use of other regular or as required medications that may affect bowel function. (e.g. codeine phosphate).
* Patients with complete or partial spinal cord injuries including cauda equina syndrome.
* Active inflammatory bowel disease.
* Pregnancy
* Stoma in situ
* Psychiatric and physiological inability to comply with study protocol.
* Non english speakers (student project funding cannot cover interpreter and other costs)

(application of criteria at the discretion of the investigating doctor at initial consultation)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
To evaluate the use of imodium as tablets or syrup in the treatment of faecal incontinence in order to improve the scores of patients with faecal incontinence as seen with continence and quality of life questionnaires | 2 sets of 6 weeks (3 months)

SECONDARY OUTCOMES:
To reduce to number of patients suffering from faecal incontinence | 3 months
Number of episodes of total, urge and passive incontinence | 3 months
Total number of patient incontinent days | 3 months
Use of pads and other medications | 3 months
Ability to defer defaecation | 3 months
Adverse effects relating to medication | 3 months
Determining the direct medical costs, direct non-medical costs, indirect non-medical costs associated with the treatment of Faecal incontinence, and cost effectiveness of treatment with syrup and tablets | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen Nugent, MA MSmedFRCS, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- Southampton General Hospital, Southampton, Hampshire, United Kingdom

REFERENCES:
- [Background] Palmer KR, Corbett CL, Holdsworth CD. Double-blind cross-over study comparing loperamide, codeine and diphenoxylate in the treatment of chronic diarrhea. Gastroenterology. 1980 Dec;79(6):1272-5. PMID 7002706
- [Background] Cheetham M, Brazzelli M, Norton C, Glazener CM. Drug treatment for faecal incontinence in adults. Cochrane Database Syst Rev. 2003;(3):CD002116. doi: 10.1002/14651858.CD002116. PMID 12917921